CLINICAL TRIAL: NCT03266666
Title: An Evaluation of Lifestyle Change Classes and Grocery Credits to Promote Healthy Behavior Change
Brief Title: Welcome to WellnessRX: Steps Toward a Healthier Life!
Acronym: WellnessRX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ProofPilot (Industry)
Collaborators: North Coast Opportunities, Inc. (Other); Thrive Market (Industry); Adventist Health Clear Lake (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 741
Record Dates: First submitted 2017-08-01; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Life Style; Behavior; Food Habits; Stress; Physical Activity
Keywords: grocery; lifestyle; lifestyle change; behavior; nutrition
MeSH Terms: conditions — Behavior; Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm - WellnessRX (Other): This is a longitudinal outcome study. All participants will receive the class and grocery credit intervention.
  Interventions: Behavioral: WellnessRX Lifestyle Change Classes; Other: Thrive Market Grocery Credits (4x$25 each)

INTERVENTIONS:
Behavioral: WellnessRX Lifestyle Change Classes — Lifestyle change classes on nutrition, physical activity, and stress management.
Other: Thrive Market Grocery Credits (4x$25 each) — Thrive Market is an online grocery service available nationwide. Participants will be provided with up to $100 on grocery credits.

SUMMARY:
Wellness Rx is a 6 class prescription for a healthier lifestyle developed for people in Lake County at all levels of health including those struggling with chronic disease. The classes are running across the community at all times. It is designed for patients that could benefit from healthy diet, exercise, and other healthy lifestyle modifications.

For those participants attending the classes, they have the option of engaging in this evaluation. For those that do, participants will answer questions about their current lifestyle, their and their previous history. They will register attendance at each class and answer questions about their perception of the class. Then at 45 days and 90 days the participants will revisit the same baseline lifestyle questionnaires.

As participants attend classes, and complete questionnaires, they'll unlock grocery credits from online food store ThriveMarket, a basket of fresh produce from the local farmers market and local fitness classes to help you towards your goals. The use of these credits will be tracked through the 90-day point.

ELIGIBILITY:
Inclusion Criteria:

* Lake County, California Resident
* able to attend 6 lifestyle change classes held around the community

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Activity Questionnaire with Eating Behaviors | 45 day
  Based on the UK National Health Service Assessments, a measure of physical activity, diet and general healthy lifestyle activities.
Activity Questionnaire with Eating Behaviors | 90 day
  Based on the UK National Health Service Assessments, a measure of physical activity, diet and general healthy lifestyle activities.
Thrive Market Purchase Decisions | through 90 days
  An analysis of purchase decisions by study participants on Thrive Market, the online natural goods store.

SECONDARY OUTCOMES:
Customer Satisfaction | within 45 minutes
  Participant perceptions of usefulness and quality of WellnessRX classes

IPD SHARING:
Plan to Share IPD: Undecided